CLINICAL TRIAL: NCT04497493
Title: Efficacy of Transcranial Direct Current Stimulation (tDCS) of Dorsolateral-prefrontal Cortex as an Add-on Treatment for Drug-naïve Major Depressive Disorder: A Randomized, Double-blind, Sham-controlled Trial
Brief Title: Efficacy of Transcranial Direct Current Stimulation (tDCS) for the Treatment of Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS-2020-TJAH
Record Dates: First submitted 2020-07-22; First posted 2020-08-04 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorders
Keywords: drug-naïve Major depressive disorder; transcranial Direct Current Stimulation (tDCS)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Experimental): participants receive 20 min sessions of 2 mA direct current delivered over the dorsolateral prefrontal cortex, 5 days per week, for 4 weeks combine a selective serotonin reuptake inhibitor (SSRI) or a serotonin and norepinephrine reuptake inhibitors(SNRI)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)-active
- Sham group (Sham Comparator): Participants receive sham stimulation that administered similarly, but with current turned off after 30s combine a selective serotonin reuptake inhibitor (SSRI) or a serotonin and norepinephrine reuptake inhibitors(SNRI)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)-sham

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS)-active — Transcranial direct current stimulation (TDC) is a non-invasive neuromodulation technique of the brain with a DC microelectrical stimulator, a cathode electrode and an anode electrode, and a control software to set the output of the stimulation type，participants receive 20 min sessions of 2 mA direct current delivered over the dorsolateral prefrontal cortex, 5 days per week, for 4 weeks
  Other Names: active
  Arms: tDCS group
Device: Transcranial Direct Current Stimulation (tDCS)-sham — Transcranial direct current stimulation (TDC) is a non-invasive neuromodulation technique of the brain with a DC microelectrical stimulator, a cathode electrode and an anode electrode, and a control software to set the output of the stimulation type. Participants receive sham stimulation over the dorsolateral prefrontal cortex, with current turned off after 30 second. The session last 20 min 5 days per week, for 4 weeks
  Other Names: sham
  Arms: Sham group

SUMMARY:
The aim of this study is to assess the efficacy of Transcranial Direct Current Stimulation (tDCS) as an Add-on Treatment for the drug-naïve Major depressive disorder. Meanwhile, evaluate the effect of tDCS on cognitive function of drug-naïve MDD patients. Furthermore, the investigators will examine the changes in cortisol, gut microbiome and some biomarkers. The hypothesis of this study is that tDCS alleviate the depressive symptoms and improve the cognitive function of drug-naïve Major depressive disorder patients with regulating inflammatory response.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled study using transcranial Direct Current Stimulation (tDCS) for 4-week treatment. After the intervention of tDCS, there is a follow up visit at week 8 in order to understand the long-term effects of tDCS. Participants were randomly assigned 1:1 to tDCS group or sham-control group. Active tDCS comprised 20 min sessions of 2 mA direct current delivered over the dorsolateral prefrontal cortex, 5 days per week, for 4 weeks. Sham was administered similarly, but with current turned off after 30s. Apart from studying the effects of tDCS on severity of depression and cognitive function, the secondary outcomes are to examine biomarkers related to inflammatory activity. Scale assessments are performed before the initiation of treatment, week 1, week 2, week 3, week 4 and week8. Collection of blood, excrement and saliva takes place at three time points, at the baseline, week 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* a current episode of MDD diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* age between 18 and 50 years
* a total score of HAMD-17 ≥ 17
* take antidepressants less than 3 days
* Patients are compliant with treatment according to the judgement of the treating clinician.

Participant or guardian has to sign informed consent. The patients' guardians will sign the informed consent on behalf of the participants when the capacity of participants to consent is compromised.

Exclusion Criteria:

* A history of manic episode
* Use of mood stabilizer
* History of substance abuse or dependence
* Severe somatic diseases that might interfere with regular antidepressant treatment including conditions such as kidney and liver failure, uncontrolled hypertension, cardiovascular, cerebrovascular and pulmonary disease, thyroid disease, diabetes, epilepsy and asthma.
* Use of anti-inflammatory medication for longer than 7 days in the last two months preceding the trial
* Use of immunosuppressive medication such as oral steroid hormones Women in pregnancy or lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The change of scores in Hamilton Depression Rating Scale (HAMD)-17 from baseline to week 4. | baseline, Week 1, week 2, week 3, week 4
  The main objective is to explore whether tDCS add on SSRI or SNRI will improve the MDD symptoms after 4 weeks of treatment, and investigators assess the scale at baseline and week 1, 2, 3, 4. Hamilton Depression Rating Scale (HAMD)-17 items was used to evaluate the severity of symptoms of depression. A total score of more than 24 may indicate severe depressive symptoms; A score above 17 may be mild to moderate depressive; If the score is less than 7, the patient has no symptoms of depression. The higher the total score of the scale, the more severe the depressive symptoms.

SECONDARY OUTCOMES:
The change of scores in Hamilton Anxiety Rating Scale (HAMA) from baseline to Week 4. | baseline, Week 1, week 2, week 3, week 4
  The aim is to explore whether tDCS add on SSRI or SNRI will alleviate the severity of anxious symptoms as measured with HAMA after 4 weeks of treatment, and investigators assess the scale at baseline and week 1, 2, 3, 4. Hamilton Anxiety Rating Scale (HAMA) was used to evaluate the severity of anxiety symptoms and the effects of intervention in patients with anxiety and depressive disorders. The total score ≥ 29 may be severe anxiety; ≥ 21, there may be obvious anxiety; ≥ 14, there may be anxiety; more than 7, there may be anxiety; if less than 7, there will be no anxiety symptoms.
The change of scores in Pittsburgh Sleep Quality Index (PSQI) from basline to week 8. | baseline, Week 4, week8
  The aim is to investigate whether active-stimuli in addition to regular treatment with an antidepressant will improve the sleep quality as measured with Pittsburgh Sleep Quality Index (PSQI) after 4 weeks of treatment compared to sham-stimuli, and investigators assess the scale at baseline and week 4,8. PSQI was used to evaluate the sleep quality of the subjects in the last month. The total score of PSQI ranged from 0 to 21. The higher the score, the worse the sleep quality.
The change of scores in quality of life (QOL) from baseline to week 8. | baseline, Week 4, week 8
  The aim is to investigate whether active-stimuli in addition to regular treatment with an antidepressant will improve the quality of life as measured with quality of life (QOL) after 4 weeks of treatment compared to sham-stimuli, and investigators assess the scale at baseline and week 4,8. The QOL scale evaluates the physical health, mental health, social relations and other aspects of the participants. The higher the score is, the better the quality of life is.
The change of sores in suicidal risk assessment scale from baseline to week 8 | baseline, Week 4, week 8
  The aim is to investigate whether active-stimuli in addition to regular treatment with an antidepressant will reduce the risk suicide as measured with the suicidal risk assessment scale after 4 weeks of treatment compared to sham-stimuli, and investigators assess the scale at baseline and week 4,8. The higher the score of the suicidal risk assessment scale, the higher the risk of suicide.
The change of scores in Repeatable Battery for the Assessment of neuropsychological Status (Rebans). | baseline, Week 4, week 8
  The aim is to observe whether active-stimuli in addition to regular treatment with an antidepressant will improve the cognitive function as measured with Repeatable Battery for the Assessment of Neuropsychological Status (Rebans) after 4 weeks of treatment compared to sham-stimuli, and investigators assess the scale at baseline and week 4,8. The higher the score of the scale, the cognitive function is better.
The changes of levels of biomarkers in peripheral blood from baseline to week 4 | baseline, week 4
  The aim is to investigate the change of cortisol level of saliva and intestinal flora as active stimuli in addition to regular treatment with an antidepressant after 4 weeks of treatment compared to sham stimuli, and investigators collect the specimens at baseline and week 4.
  Saliva collection tube to collect saliva, collect naturally discharged saliva in a clean test tube (at least 2ml). Saliva was centrifuged under 1500rpm for 15 minutes and the filtrate was cryopreserved at-80 °C. the saliva was analyzed by ELISA kit.
  Fecal collection: a) intercept the middle part of the sample with a sterile toothpick or fecal sampler (the surface of feces contains exfoliated cells of intestinal mucosa; the outside is easy to be contaminated, and some bacterial DNA begins to degrade after contact with air), take about the size of peanuts and put them into aseptic 2.0mL centrifuge tubes, 3-5 tubes for each sample are taken for backup，and then put into-80 °C cryopreservation after sub-packaging.
Adverse events from baseline to week 4 | week 1, week 2, week 3, week 4
  The aim is to evaluate the adverse effects during the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided